CLINICAL TRIAL: NCT06424366
Title: ADAPT: Approach to Dance for Autism
Brief Title: Approach to Dance for Autism
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: American Psychiatric Association (Other)
Responsible Party: Principal Investigator, Alexander Kolevzon, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00144
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Ballet; Autism; Motor; Recreational; Children; Dance
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The study will use a waitlist control design. The first arm will be the experimental arm and will immediately begin the intervention post recruitment. The second arm will be the waitlist control arm and will begin the intervention after the first arm's completion.
Masking Description: Due to the nature of the intervention (ballet classes) and that caregivers will be completing all questionnaires, masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Ballet Program (Experimental): 12 weeks of ballet classes immediately after recruitment and randomization concludes.
  Interventions: Behavioral: Ballet for All Kids
- Deferred Ballet Program (Placebo Comparator): 12 weeks of ballet classes after the first arm completes the intervention. Participants in this arm will continue to complete self-reports while they wait to begin the intervention.
  Interventions: Behavioral: Ballet for All Kids

INTERVENTIONS:
Behavioral: Ballet for All Kids — The intervention consists of 12 weeks of ballet classes that follow the structure and curriculum of Ballet for All Kids (BFAK). BFAK is a non-profit organization that has been tailoring ballet classes for children with autism spectrum disorder for over one decade. Ballet classes will be held once a week for 45 minute sessions and led by trained medical and graduate students who have successfully completed BFAK's training and certification. BFAK instruction is based on the Schlachte Method, which combines auditory, visual, vestibular, and emotional learning to individualize instruction to match each child's skill level. In classroom accommodations include, but are not limited to a visual schedule, personal dance areas demarcated by tape on the floor, and one-on-one volunteer assistance.

SUMMARY:
This study will be a randomized trial that will examine the impact of a recreational ballet program on children with autism spectrum disorder (ASD). The research team are primarily interested in assessing changes in motor skills with secondary objectives focused on the social, psychological, and behavioral effects. The study will aim to collect data from 24 participants with ASD. Participants must be 7-12 years old, have a confirmed diagnosis of ASD, and speak English or Spanish. All participants will be enrolled in a 12 week ballet program. The ballet program is based off the curriculum and structure of Ballet for All Kids, a non-profit organization that has been tailoring ballet classes for children with ASD for over one decade. All research team members and volunteers will be trained in the BFAK program's curriculum and structure. Ballet instruction and all research materials will be provided in both English and Spanish. The research team will randomize the sample into an intervention group and waitlist control. The research team will measure outcomes through validated self-reports that caregivers will complete. For the intervention group, questionnaires will be completed at baseline and throughout the intervention (weeks 4, 8, and 12). For those in the waitlist control group, questionnaires will be completed at baseline, throughout the intervention group's ballet classes, and throughout their own participation in the program. Results of this study will help to determine if how a recreational ballet program can impact the motor, psychological, social, and behavioral skills of a child with ASD, informing the direction of future research and interventions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autism spectrum disorder
* Fluent in English or Spanish
* Between 7-12 years old

Exclusion Criteria:

* For any reason the individual appears unable to participate in study procedures per the Principal Investigator
* Not fluent in English or Spanish
* Unable to commit to at least 8 of the 12 scheduled intervention sessions

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Development Coordination Disorder Questionnaire | at baseline and weeks 4, 8, and 12
  Development Coordination Disorder Questionnaire will be completed by caregivers and will assess participants' motor skills throughout the study. Minimum score= 15. Maximum score= 75. A higher score indicates more advanced motor skills.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist | at baseline and weeks 4, 8, and 12
  The Aberrant Behavior Checklist will be completed by caregivers and will assess participants' behaviors such as irritability; lethargy; stereotypy; hyperactivity; and inappropriate speech. Minimum score= 0. Maximum score= 174. A higher score indicates a greater degree of that behavior (i.e. higher scores on irritability would indicate that child tends to be more irritable).
Social Responsiveness Scale 2 | at baseline and weeks 4, 8, and 12
  The Social Responsiveness Scale 2 will be completed by caregivers and will assess participants' social behaviors throughout the study. Minimum raw score = 65. Maximum raw score = 260. T-scores have a mean of 50 and a SD of 10. Raw scores are converted to T scores based on the child's gender. A higher score indicates more severe social impairments.
Children's Sleep Habits Questionnaire (Abbreviated) | at baseline and weeks 4, 8, and 12
  The Children's Sleep Habits Questionnaire will be completed by caregivers and will assess participants' sleep throughout the study. Minimum score = 0. Maximum score = 154. A higher score indicates more sleep disturbances.
The Repetitive Behavior Scale | at baseline and weeks 4, 8, and 12
  The Repetitive Behavior Scale will be completed by caregivers and will assess participants' repetitive behaviors and restricted interests throughout the study. Minimum score = 0. Maximum score = 129. A higher score indicates more severe behaviors.
Caregiver Strain Questionnaire | at baseline and weeks 4, 8, and 12
  The Caregiver Strain Questionnaire will be completed by caregivers and will assess caregivers' stress related to parental/familial responsibilities throughout the study. Minimum score = 21. Maximum score = 105. A higher score indicates that a caregiver experiences more distress due to their familial responsibilities.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size, recruitment of minor populations, and sensitive nature of some of the questionnaires, we will not be sharing IPD.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT06424366/ICF_000.pdf